CLINICAL TRIAL: NCT04868292
Title: A Phase 1, Single-Center, Open-Label Study to Assess the Intrapulmonary Pharmacokinetics of SPR206 by Comparing the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations Following the Intravenous Administration of SPR206 in Healthy Volunteers
Brief Title: Study to Assess the Intrapulmonary Pharmacokinetics of SPR206 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPR206-102; CDMRP-JW180095-A (Other Grant/Funding Number: United States Department of Defense); 2020-006019-52 (EudraCT Number)
Record Dates: First submitted 2021-04-13; First posted 2021-04-30 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; alveolar macrophages (AM); epithelial lining fluid (ELF); intrapulmonary; bronchoalveolar lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPR206 (Experimental): Healthy subjects meeting eligibility criteria will receive a total of three 100 mg SPR206 intravenous doses administered every 8 hours.
  Interventions: Drug: SPR206

INTERVENTIONS:
Drug: SPR206 — Three 100 mg SPR206 intravenous doses administered every 8 hours

SUMMARY:
To evaluate the intrapulmonary pharmacokinetics (PK), including epithelial lining fluid (ELF) and alveolar macrophage (AM) concentrations, of SPR206 as well as plasma concentrations of SPR206 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker for at least 12 months prior to screening for the study
* BMI ≥ 18.5 and ≤ 32 (kg/m2) and weight between 55.0 and 100.0 kg (both inclusive)
* Medically healthy without clinically significant abnormalities as assessed by the Investigator based on screening medical history, physical examination, vital signs, 12-lead ECG, hematology, biochemistry, coagulation, and urinalysis
* Forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value at screening
* Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food from 48 hours prior to study drug administration until discharge from the clinical unit
* If male, must agree to use a condom and have a non-pregnant female partner of childbearing potential agree to use a highly effective method of contraception
* If female, must be of non-childbearing potential or, if female of childbearing potential, a willingness to abstain from sexual activity or agree to use a high effective method of contraception that could lead to pregnancy
* Other inclusion criteria per protocol

Exclusion Criteria:

* History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, vascular or neurological disease, including any acute illness or surgery within the past 3 months determined by the Investigator to be clinically relevant
* Recent history (within 6 months) of known or suspected Clostridium difficile infection
* History of seizure disorders
* Positive urine drug, alcohol or cotinine testing at screening or check-in (Day -1)
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV Ab)
* Positive testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening or prior to first dosing
* Presence of the following symptoms at screening or within 28 days prior to screening or check-in (Day -1):

  1. Fever, chills or sweats (temperature of 38 °C / 100.4 °F or higher)
  2. Difficulty breathing
  3. Cough
  4. Sore throat
  5. New or recent loss of taste or smell
  6. Nausea, vomiting or diarrhea
* Close contact with anyone who tested positive for SARS-CoV-2 infection within 28 days prior to screening or check-in (Day -1)
* Electrocardiogram (ECG) with QTcF interval duration equal or greater than 450 msec for males and 470 msec for females
* Subjects who have any of the following abnormalities on laboratory values at screening or Check-In including:

  1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL
  2. Absolute neutrophil count ≤ 2,000/mm3, platelet count <120,000/mm3
  3. alanine aminotransferase (ALT) OR aspartate aminotransferase (AST) greater than the upper limit of normal (ULN) for the reference laboratory
* History of substance abuse or alcohol abuse
* Use of prescription medicine & tobacco/nicotine or marijuana-containing products
* A female who is pregnant or breastfeeding
* Other exclusion criteria per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to 8 hours (AUC0-8) for ELF, AM, and plasma | 8 hours after the start of the third study drug IV infusion
Maximum observed concentration (Cmax) for ELF, AM, and plasma | 8 hours after the start of the third study drug IV infusion
Minimum concentration (Cmin) for ELF, AM, and plasma | 8 hours after the start of the third study drug IV infusion
Time to the maximum observed concentration (Tmax) for ELF, AM, and plasma | 8 hours after the start of the third study drug IV infusion

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day -1 to Day 7
  To assess the incidents of treatment-emergent adverse events following three 100mg SPR206 intravenous doses administered every 8 hours. AEs will be classified by System Organ Class (SOC) and Preferred Term (PT). Incidence, frequency, severity and duration will be presented.
Incidence of abnormal vital sign assessments - blood pressure | Day -1 to Day 7
  To assess the incidents of abnormal systolic and diastolic blood pressure assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Frequency count of significant changes from baseline will be presented.
Incidence of abnormal vital sign assessments - body temperature | Day -1 to Day 7
  To assess the incidents of abnormal body temperature assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Frequency count of significant changes from baseline will be presented.
Incidence of abnormal vital sign assessments - heart rate | Day -1 to Day 7
  To assess the incidents of abnormal heart rate assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Frequency count of significant changes from baseline will be presented.
Incidence of abnormal vital sign assessments - respiratory rate | Day -1 to Day 7
  To assess the incidents of abnormal respiratory rate assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Frequency count of significant changes from baseline will be presented.
Incidence of abnormal physical exam assessments | Day -1 to Day 7
  To assess the incidents of abnormal body system assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Changes from baseline in physical examination findings will be classified as Normal, Abnormal NCS, and Abnormal CS. Frequency counts will be presented.
Incidence of abnormal ECG assessments - heart rate | Day -1 to Day 7
  To assess the incidents of abnormal heart rate assessment following three 100mg SPR206 intravenous doses administered every 8 hours. Cardiac (12-Lead ECG) for heart rate will be classified as normal, abnormality that is NCS, and CS abnormality. Frequency counts by dose group and timepoint of collection will be presented.
Incidence of abnormal ECG assessments - PR, RR, QRS, QT and QTcF interval | Day -1 to Day 7
  To assess the incidents of abnormal PR interval, RR interval, QRS interval, QT interval and QTcF interval assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Cardiac (12-Lead ECG) results will be classified as normal, abnormality that is NCS, and CS abnormality. Frequency counts by dose group and timepoint of collection will be presented.
Incidence of abnormal safety laboratory assessments | Day -1 to Day 7
  To assess the incidents of abnormal hematology, serum chemistry, coagulation and urinalysis assessments following three 100mg SPR206 intravenous doses administered every 8 hours. Frequency counts of significant changes from baseline will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — Spero Therapeutics Inc
Locations (1):
- Medical Facility, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No